CLINICAL TRIAL: NCT01619865
Title: Safety & Efficacy of 68Ga-DOTA-tyr3-Octreotide PET/CT in Diagnosis, Staging & Measurement of Response to Treatment in Patients With Somatostatin Receptor Positive Tumors: Comparison to Octreoscan Plus High-Resolution, Contrast Enhanced CT.
Brief Title: Safety of 68Ga-DOTA-tyr3-Octreotide PET in Diagnosis of Solid Tumors
Acronym: GA-68
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sue O'Dorisio (Other)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201110718; 114398 (Other: FDA)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumors; Neuroblastoma; Medulloblastoma
Keywords: GA-68; Gallium 68; GA-68 PET
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Neuroblastoma; Medulloblastoma | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Masking Description: The Octreoscan and 68Ga-DOTA-tyr3-Octreotide PET scans are read independently by two certified nuclear medicine physicians for discordant positive lesions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATOC PET/CT (Experimental): 68Ga-DOTATOC Positron Emission Tomography (PET) for Diagnosis, Staging, and Measurement of Response to Treatment in Somatostatin Receptor Positive Tumors
  Interventions: Drug: 68Ga-DOTATOC PET/CT

INTERVENTIONS:
Drug: 68Ga-DOTATOC PET/CT — 1 -5 mCi 68Ga-DOTATOC (10-50 ugm DOTATOC)administered once via IV.
  Other Names: Gallium 68-DOTATOC

SUMMARY:
This protocol is designed to test the efficacy of 68Ga-DOTATOC PET/CT in diagnosis, staging, and measurement of response to treatment in patients with somatostatin receptor positive tumors. Goals are to 1) compare this unique PET/CT scan with the current standard of care which is a combination of Octreoscan SPECT (single photon emission tomography) plus a high resolution, contrast enhanced CT; 2) Determine the sensitivity of 68Ga-DOTATOC PET/CT in diagnosis of patients with suspected somatostatin receptor positive tumor; and 3) For those patients who have had recent treatment (e.g., surgery, chemotherapy, targeted therapy such as anti-angiogenics, kinase inhibitors, peptide receptor radiotherapy), this scan will be used to measure response to treatment. These studies will be obtained with the long term goal of submitting a New Drug Application (NDA) for FDA approval of 68Ga-DOTATOC PET/CT in adults and children.

DETAILED DESCRIPTION:
This protocol is designed to test the efficacy of 68Ga-DOTATOC PET/CT in diagnosis, staging, and measurement of response to treatment in patients with somatostatin receptor positive tumors. The goals are to 1) compare this unique PET/CT scan with the current standard of care which is a combination of Octreoscan SPECT (single photon emission tomography) plus a high resolution, contrast enhanced CT; 2) Determine the sensitivity of 68Ga-DOTATOC PET/CT in diagnosis of patients with suspected somatostatin receptor positive tumor; and 3) For those patients who have had recent treatment (e.g., surgery, chemotherapy, targeted therapy such as anti-angiogenics, kinase inhibitors, peptide receptor radiotherapy), this scan will be used to measure response to treatment. These studies will be obtained with the long term goal of submitting a New Drug Application (NDA) for FDA approval of 68Ga-DOTATOC PET/CT in adults and children.

Project Design

68Ga-DOTATOC Positron Emission Tomography (PET) for Diagnosis, Staging, and Measurement of Response to Treatment in Somatostatin Receptor Positive Tumors is a prospective, Phase 1-2, single center, open-label study in subjects with known or suspected somatostatin receptor positive tumor. Eligible participants will undergo baseline assessments at enrollment. Study participants will receive 68Ga-DOTATOC and undergo a PET/CT imaging study with an option to receive a second 68Ga-DOTATOC PET/CT if they begin a new treatment (surgery, hepatic embolization, Sandostatin LAR, chemotherapy, targeted biological therapy, or peptide receptor radiotherapy) within 30 days of the first scan. The second scan will be performed at a time recommended by the treating physician as optimal interval to observe results from treatment.

Project Goal

This study is planned to demonstrate the safety and efficacy of [68Ga]-DOTA-tyr3-Octreotide ([68Ga]-DOTATOC) as an accurate imaging technique for diagnosis, staging, and monitoring of response to treatment in patients with Somatostatin receptor expressing tumors.

Neuroendocrine tumors are solid malignant tumors that arise from dispersed neuroendocrine cells found throughout the body. Gastroenteropancreatic neuroendocrine tumors (NETs) can be divided into two groups: Carcinoid tumors that may arise from the lungs, stomach, small bowel or colon and pancreatic neuroendocrine tumors (also known as pancreatic islet cell tumors). The clinical behavior of NETs is extremely variable; some may cause hormone hypersecretion and others may not, the majority of them are slow-growing tumors (well-differentiated NETs), whereas some NETs are highly aggressive (poorly differentiated NETs). The incidence of NETs is increasing, from 1.1/100,000 per year in 1973 to 5.3/100,000 per year in 20041. Among NETs, 25% have distant metastases and 25% have regional involvement at the time of initial diagnosis[1]. Other tumors that express high levels of somatostatin receptors include neuroblastoma, medulloblastoma, and Ewing's sarcoma[2-4].

The radiological detection and staging of these tumors is challenging and requires a multimodality approach. Somatostatin receptor imaging with In-111 Pentetreotide (OctreoScan) and multiphase CT are the most commonly used modalities although the use of endoscopic ultrasound and MRI is also increasing. Surgery is the only curative option for NETs. However, curative surgery in malignant NET is possible in less than 30% of patients with recurrence identified in the majority of patients as late as 15 years after initial surgery. Treatment with somatostatin analogs, which include the short acting subcutaneous and long acting release (LAR) octreotide, are effective in stabilizing NETs and have been recently demonstrated to prolong the time to progression of disease[5]. Chemotherapy is generally not effective in low grade NETs, but it may be helpful in high grade and pancreatic NETs. On the other hand, neuroblastoma, medulloblastoma, and Ewing's sarcoma are initially responsive to chemotherapy, but relapses are common and salvage therapies are not very effective, resulting in <30% overall survival at 5 years[6-8].

Somatostatin Receptor Targeted Imaging and Therapy

Tumors that express somatostatin receptors can be targeted with radiolabeled somatostatin analogues for imaging and treatment. Somatostatin receptor gamma camera imaging with In-111 DTPA-octreotide (OctreoScan) targeting somatostatin receptor 2 (sstr2), is used routinely for imaging of neuroendocrine tumors with a detection rate >90% for well-differentiated carcinoid tumors and majority of pancreatic NETs, but only a 50% detection rate for insulinomas, which may show a weaker expression of sstr2[9].

Given the clinical efficacy of this radiolabeled peptide as a diagnostic agent, studies to test if therapeutic radiation could be targeted to tumors in a similar manner was a logical next step. Attempts to utilize In-111 DTPA Octreotide as a therapeutic agent have been minimally effective due to short range of auger electrons utilized in this therapy. The efficacy of this treatment was improved with the development of somatostatin analogues labeled with beta emitting radioisotopes. Further studies have identified DOTA as a superior chelator compared to DTPA, increasing the stability and receptor targeting of somatostatin analogues[10]. There is now a large clinical experience with Yttrium-90 DOTA-tyr3-Octreotide peptide radioreceptor therapy (PRRT) in Europe, primarily in adults with neuroendocrine tumors[11]. An international Phase II clinical trial then followed and included several trial sites in the United States, notably the University of Iowa, where we entered 40 subjects[12]. With its low toxicity profile, the significant improvement in symptoms and quality of life and the lack of effective alternative therapies, PRRT has been suggested as possible first-line therapy in adult patients with gastroenteropancreatic neuroendocrine tumor. Recent data have also demonstrated a significant survival benefit with PRRT compared to historical controls in this population. We have also now conducted a Phase I trial of 90Y-DOTA-tyr3-Octreotide in children and young adults at the University of Iowa, which also shows promise of efficacy of this treatment in pediatric patient population[13]. We now propose a new imaging agent for use in diagnosis and therapy of Somatostatin receptor positive tumors.

Somatostatin Receptor PET Imaging with Ga-68 DOTA0-Tyr3-octreotide

More recently, positron emission tomography (PET) radiopharmaceuticals have been developed that can be labeled with Gallium-68 (Ga-68). Gallium-68 is a generator product with a half-life of 68 min (compared to 67 hours for In-111 in OctreoScan). The parent nuclide of Ga-68 is Germanium-68, which has a half-life of 270.8 days. Ga-68 decays by 89% through positron emission and 11% by electron capture. Its parent, A number of Ga-68 DOTA-conjugated peptides have been introduced, including Ga-68 DOTA0-Tyr3]octreotide (Ga-68 DOTATOC), Ga-68 DOTA0-1NaI3-octreotide (Ga-68 DOTANOC) and [Ga-68 DOTA0-Tyr3]octreotate (Ga-68 DOTATOC). All of these radiolabeled peptides bind to sstr2, although DOTANOC also binds to sstr 3 and sstr 5, and DOTATOC to sstr5[14]. The primary advantage of Ga-68 based somatostatin receptor PET imaging over OctreoScan SPECT is the higher imaging resolution and accurate quantitation of uptake due to robust attenuation correction. The improved resolution and quantitation of uptake obtained with Ga-68 DOTATOC PET should provide a more accurate assessment of somatostatin receptor density, which will lead to a more accurate prediction of treatment response to somatostatin analogues. A recent study from Europe comparing Ga-68 DOTATOC with Octreoscan found Ga-68 DOTATOC to be superior in detection of skeletal and pulmonary involvement of neuroendocrine tumors[15].

Rationale and overall study design

Rationale:68Ga-DOTATOC positron emission tomography (PET) scanning and 90Y-DOTATOC peptide receptor radionuclide therapy (PRRT) are readily available in Europe, but neither radiopharmaceutical is approved for use in the United States. IND #61,907 is currently active under the above named investigators for 90Y-DOTATOC PRRT in somatostatin receptor positive tumors. These investigators have conducted a single institution Phase I trial of 90Y-DOTATOC therapy in children and young adults (Appendix I) and have participated in a Phase II trial of 90Y-DOTATOC PRRT in adults (also in Appendix II).

The purpose of this amendment to the IND application is to test the efficacy of 68Gallium-DOTATOC in diagnosis, staging, and determination of response to 90Y-DOTATOC PRRT in children and adults with known or suspected somatostatin receptor positive tumors, including, but not limited to neuroendocrine tumors, neuroblastoma, and medulloblastoma. 68Ga-DOTATOC PET would replace 111In-DTPA-Octreotide single photon emission tomography (SPECT) imaging. Whereas, Octreoscan uses a 222 MBq imaging dose of Indium (2.8 day half life) resulting in an effective dose equivalent (HE) equal to 2.61 rads, [68Ga]DOTATOC (68 min half life) uses 185 MBq with an effective dose equivalent of 0.46 rads. In addition, [68Ga]DOTATOC PET/CT can be completed within 2 hours compared to an Octreoscan which requires 3 visits over 24 hours, making [68Ga]DOTATOC a much more convenient imaging choice for patients. The data obtained in this Ga-68 DOTATOC PET study will be used to support the use of 68Ga-DOTATOC PET for diagnosis and staging in patients with suspected or proven somatostatin receptor positive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age greater than or equal to 2 years
* Known or suspected somatostatin receptor positive tumor such as carcinoid; neuroendocrine tumor; neuroblastoma; medulloblastoma; pheochromocytoma. Supporting evidence may include MRI, CT, biochemical markers, and or pathology report.
* Karnofsky performance status or Lansky Play Scale status of greater than 50 (or ECOG/WHO equivalent)
* Subject is male; or is a female who is either pre-menarchal, surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (> 1 years without menses), non-lactating, or of childbearing potential for whom a serum pregnancy test (with the results known prior to investigational product administration) is negative. A negative serum pregnancy test will be required for all female subjects with child bearing potential. If a false pregnancy test is suspected, e.g., perimenopausal condition, an obstetrician will be consulted to determine if she is/is capable of becoming pregnant.

Exclusion Criteria:

* Subject weighs more than 400 pounds (Subjects who weigh more than 400 pounds will not be able to fit inside the imaging machines).
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.)
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Does the subject have any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance?

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2017-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue O'Dorisio, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD are entered into the subject's electronic medical record and are shared with referring physicians when obtained.
Supporting Information: CSR
Time Frame: Results are shared when clinically available.
Access Criteria: Results are placed in patient's electronic medical record.

REFERENCES:
- [Result] Abongwa C, Mott S, Schafer B, McNeely P, Abusin G, O'Dorisio T, Zamba G, O'Dorisio MS, Menda Y. Safety and accuracy of 68Ga-DOTATOC PET/CT in children and young adults with solid tumors. Am J Nucl Med Mol Imaging. 2017 Nov 1;7(5):228-235. eCollection 2017. PMID 29181270
- [Result] Menda Y, O'Dorisio TM, Howe JR, Schultz M, Dillon JS, Dick D, Watkins GL, Ginader T, Bushnell DL, Sunderland JJ, Zamba GKD, Graham M, O'Dorisio MS. Localization of Unknown Primary Site with 68Ga-DOTATOC PET/CT in Patients with Metastatic Neuroendocrine Tumor. J Nucl Med. 2017 Jul;58(7):1054-1057. doi: 10.2967/jnumed.116.180984. Epub 2017 Feb 2. PMID 28153957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Iowa Holden Comprehensive Cancer Center Clinics and University of Iowa Children's Hospital. Participants being seen for known or suspected somatostatin receptor positive tumors were recruited for the study. Malignancies included neuroblastoma, medulloblastoma, and pheochromocytoma.
Pre-assignment Details: Female subjects of childbearing potential were given a pregnancy test (serum) prior to receiving research-related radiation. A women who was pregnant could not participate in the study.
Groups:
- 68Ga-DOTATOC PET/CT: 68Ga-DOTATOC Positron Emission Tomography (PET) for Diagnosis, Staging, and Measurement of Response to Treatment in Somatostatin Receptor Positive Tumors
  68Ga-DOTATOC PET/C: 1 -5 mCi 68Ga-DOTATOC (10-50 ugm DOTATOC)administered once via IV.
Period: Overall Study
Arm/Group | 68Ga-DOTATOC PET/CT
Started | 223
Completed | 219
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — subject not able to comply | 1

BASELINE CHARACTERISTICS:
Population: Subjects with known neuroendocrine tumor with lesion identified on CT or MRI. Subjects with suspected neuroendocrine tumor with no lesion identified on CT or MRI.
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 32
  >=65 years | 182
Age, Continuous [Mean (Full Range); unit: years] | 53 [3 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 215
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 209
  More than one race | 1
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 223

OUTCOME MEASURES:

1. Primary Outcome: To Measure Safety of 68Ga-DOTATOC Positron Emission Tomography (PET) by Measuring the Number of Adverse Events Related to the Investigational Radiopharmaceutical Agent
Description: Subject receives an injection of 68Ga-DOTATOC, a somatostatin-like peptide that binds to somatostatin receptor and is tagged with a radionuclide that can be detected by positron emission tomography (PET). Whole body PET is performed; patient is queried regarding any adverse events immediately and again 24 hrs after completion of scan read by certified nuclear medicine physician to determine if any known tumor lesions take up 68Ga-DOTATOC.Severity of adverse events will be graded according to NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0). Adverse events are assessed immediately after PET scan and 24 hrs after completion of the scan.
Time Frame: During PET scan and 24 hours post scan
Population: Subjects who reported an adverse event and relationship of adverse event to study drug (68Ga-DOTATOC). Several subjects reported more than one adverse event; thus, the number of subjects who experienced an event will be less than the number of events.
Measure: Number; unit: Adverse events reported
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 105
Adverse events reported
  Possibly related | 18
  Probably related | 1
  Unlikely related | 6
  Unrelated | 157

2. Primary Outcome: Number of Subjects With Adverse Events Related to the Use of the 68Ga-DOTATOC
Description: Number of subjects with adverse events related to the use of the 68Ga-DOTATOC radiopharmaceutical in accordance with National Cancer Institute (NCI) toxicity guidelines (NCI Common Terminology Criteria for Adverse Events version 4.0)
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATOC PET/CT
Number analyzed (Participants) | 223
Participants
  Number of subjects with no adverse events (AE) | 118
  Number of subjects with Grade 1 or 2 AE | 101
  Number of subjects with Grade 3 AE | 4
  Number of subjects with Grade 4 or 5 AE | 0

ADVERSE EVENTS:
Time Frame: From time of study drug injection, through PET scan up to 24 hours post injection.
Arm/Group | 68Ga-DOTATOC PET/CT
All-Cause Mortality (participants affected / at risk) | 2/223
Serious Adverse Events (participants affected / at risk) | 1/223
Other Adverse Events (participants affected / at risk) | 176/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-DOTATOC PET/CT (N=223)
Nausea (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized of specific area (not due to neuropathy - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain NOS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-DOTATOC PET/CT (N=223)
Hemoglobin (Hepatobiliary disorders) | 12 (12)
Leukocytes (total WBC) (Hepatobiliary disorders) | 4 (4)
Lymphopenia (Hepatobiliary disorders) | 11 (11)
Platelets (Hepatobiliary disorders) | 2 (2)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 (1) — palpatations
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Sweating (diaphoresis) (General disorders) | 7 (7)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3 (3)
Flushing (Skin and subcutaneous tissue disorders) | 6 (6)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, __) (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 4 (5)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (7)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 13 (13)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 5 (5)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 5 (5)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 2 (2)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Pain - Abdomen NOS (Musculoskeletal and connective tissue disorders) | 11 (13)
Pain - Back (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain - Head/headache (Nervous system disorders) | 4 (4)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Other (Specify, __) (General disorders) | 1 (1)
Pain - Throat/pharynx/larynx (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 1 (1)
Pain-neck (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT01619865/Prot_SAP_000.pdf